CLINICAL TRIAL: NCT05254743
Title: A Phase 3 Open-Label, Randomized Study of Pirtobrutinib (LOXO-305) Versus Ibrutinib in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (BRUIN-CLL-314)
Brief Title: A Study of Pirtobrutinib (LOXO-305) Versus Ibrutinib in Participants With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Acronym: BRUIN-CLL-314
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18281; J2N-OX-JZNU (Other: Eli Lilly and Company); LOXO-BTK-20030 (Other: Eli Lilly and Company); 2023-507699-38-00 (EU CTIS Number)
Expanded Access: NCT05172700 (Approved for marketing)
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia, Lymphocytic; Leukemia, B-cell; Small Lymphocytic Lymphoma
Keywords: BTKi; Hematologic Disease; Lymphoma, non-Hodgkin's; Lymphoma, B-cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Lymphoid; Leukemia, B-Cell; Hematologic Diseases; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — pirtobrutinib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pirtobrutinib Part 1 (Experimental): Participants will receive pirtobrutinib orally.
  Interventions: Drug: Pirtobrutinib
- Ibrutinib (Active Comparator): Participants will receive ibrutinib orally.
  Interventions: Drug: Ibrutinib
- Pirtobrutinib Part 2 (Experimental): Participants will receive pirtobrutinib orally.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally.
  Other Names: LOXO-305; LY3527727
  Arms: Pirtobrutinib Part 1; Pirtobrutinib Part 2
Drug: Ibrutinib — Administered orally.
  Arms: Ibrutinib

SUMMARY:
The purpose of Part 1 of this study is to compare the efficacy and safety of pirtobruitinib (LOXO-305) to ibrutinib in participants with CLL/SLL; participants may or may not have already had treatment for their cancer. The purpose of Part 2 of this study evaluates pirtobrutinib monotherapy in treatment-naïve participants with CLL/SLL with 17p deletions. Participation could last up to six years for Part 1. Participation could last up to 2 years for Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL/SLL requiring therapy per iwCLL 2018 criteria
* Part 1 - Known 17p deletion status (wildtype or deleted). Part 2 - Must have deletion of 17p as determined by FISH testing
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Adequate organ function

  * Platelets greater than or equal to ≥ 50 x 10⁹/liter (L) or ≥30 x 10⁹/L in participants with documented bone marrow involvement considered to impair hematopoiesis,
  * Hemoglobin ≥8 grams/deciliter (g/dL) or ≥6 g/dL in participants with documented bone marrow involvement considered to impair hematopoiesis
  * Absolute neutrophil count ≥0.75 x 10⁹/L or ≥0.50 × 10⁹/L in participants with documented bone marrow involvement considered to impair hematopoiesis
  * Kidney function: Estimated creatinine clearance ≥30 milliliters per minute (mL/min)

Exclusion Criteria:

* Known or suspected Richter's transformation to diffuse large B-cell lymphoma (DLBCL), prolymphocytic leukemia, or Hodgkin's lymphoma at any time preceding enrollment
* Known or suspected central nervous system (CNS) involvement
* A significant history of renal, neurologic, psychiatric, endocrine, metabolic or immunologic disease
* Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP])
* Significant cardiovascular disease including ejection fraction < 40% and any grade ongoing atrial fibrillation or atrial flutter
* Hepatitis B or hepatitis C testing indicating active/ongoing infection, based on Screening laboratory tests
* Active cytomegalovirus (CMV) infection
* Active uncontrolled systemic bacterial, viral, or fungal infection
* Known human immunodeficiency virus (HIV) infection, regardless of cluster of differentiation 4 (CD4) count
* Clinically significant active malabsorption syndrome or other condition likely to affect GI absorption of the oral-administered study treatments
* Ongoing inflammatory bowel disease
* Previous treatment for CLL/SLL - Part 1: Treatment-naïve and previously treated, except prior exposure to BTK inhibitor (covalent or noncovalent).

Part 2: participants must be treatment naïve

* Concurrent use of investigational agent or anticancer therapy except hormonal therapy
* Participants requiring therapeutic anticoagulation with warfarin or another Vitamin K antagonist
* Use of > 20 mg prednisone daily or equivalent dose of steroid at the time of first dose of study drug
* Vaccination with a live vaccine within 28 days prior to randomization
* Participants receiving chronic therapy with a strong cytochrome P450 (CYP)3A inhibitor (except posaconazole and voriconazole) which cannot be stopped within 3-5 half lives of the CYP3A inhibitor therapy prior to start of study drug treatment
* Participants with known hypersensitivity, including anaphylaxis, to any component or excipient of pirtobrutinib or ibrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Complete Response (CR), Complete Remission with Incomplete Hematologic Recovery (Cri), Nodular Partial Remission (nPR) or Partial Response (PR): Overall Response Rate (ORR) Part 1 | Baseline to best overall response the best response recorded from Cycle 1 Day 1 until data cutoff date, PD, or start of new anticancer treatment, whichever is the earliest] (approximately 3 years and 5 months)
  ORR as assessed by independent review committee (IRC) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria
Percentage of Participants Achieving Complete Response (CR), Complete Remission with Incomplete Hematologic Recovery (CRi), Nodular Partial Remission (nPR) or Partial Response (PR): Overall Response Rate (ORR) Part 2 | Baseline to best overall response the best response recorded from Cycle 1 Day 1 until data cutoff date, PD, or start of new anticancer treatment, whichever is the earliest (Approximately 2 years and 3 months)
  ORR as assessed by independent review committee (IRC) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria

SECONDARY OUTCOMES:
IRC-assessed Progression-Free Survival (PFS) | Randomization to PD (per iwCLL 2018 criteria) or death from any cause (approximately 5 years 8 months)
  PFS by IRC per iwCLL 2018 criteria
Investigator assessed Progression-Free Survival (PFS) | Randomization to PD (per iwCLL 2018 criteria) or death from any cause (approximately 5 years 8 months)
  PFS by Investigator per iwCLL 2018 criteria
Event-Free Survival (EFS) | Randomization to first occurrence of treatment discontinuation due to adverse event/toxicity, treatment-emergent atrial fibrillation or atrial flutter of any grade, progressive disease (PD) or death (approximately 4 years)
  EFS by IRC per iwCLL 2018 criteria
Duration of Response (DOR) | Time from the date of the first documented response of CR, CRi, nPR or PR to the earlier of documentation of definitive PD (per iwCLL 2018 criteria) or death from any cause (approximately 2 years)
  DOR by IRC and Investigator by iwCLL 2018 Criteria.
Overall Survival (OS) | Randomization to death from any cause (approximately 6 years)
  OS
Time to Next Treatment (TTNT) | Randomization to initiation of the next systemic anticancer therapy for CLL/SLL or death from any cause, whichever occurs first (approximately 6 years)
  TTNT
Time to Worsening (TTW) of CLL/SLL Related Symptoms | Randomization to time to worsening symptoms (approximately 4 years)
  Using symptom questions identified from the EORTC item library. The range of raw scores for these items could be from 0 to 52 with highest score being worse symptoms.
Comparative Tolerability | From Baseline to Treatment Discontinuation for Any Reason (approximately 4 years)
  Comparative Tolerability measured by proportion of time with high side-effect burden
Percentage of Participants Achieving DOR Part 2 | Time from the date of the first documented response of CR, CRi, nPR, or PR to the earlier of the documentation of definitive PD or death from any cause] (Approximately 2 years)
  DOR as assessed by IRC and Investigator defined as the time from the date of the first documented response of CR, CRi, nPR, or PR to the earlier of the documentation of definitive PD per iwCLL 2018 criteria or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (144):
- United States (19):
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - TOI Clinical Research, Cerritos, California
  - Stanford School of Medicine-Cancer Clinical Trials Office, Palo Alto, California
  - California Cancer Associates for Research and Excellence, San Marcos, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Cancer Specialists of North Florida -St Augustine, Saint Augustine, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Tulane Cancer Center Office of Clinical Research, New Orleans, Louisiana
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Cancer Care Associates of York, York, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Kelsey Research Foundation, Houston, Texas
  - Lumi Research, Kingwood, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Medical Oncology Associates, PS, Spokane, Washington
  - MultiCare Health System Institute for Research and Innovation, Spokane, Washington
- Argentina (3):
  - Alexander Fleming, Ciudad Autónoma de Buenos Aire
  - Hospital Privado De Comunidad, Mar del Plata
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares, Santa Fe
- Australia (3):
  - One Clinical Research, Nedlands
  - Western Health, Sunshine Hospital, St Albans
  - The Perth Blood Institute, West Perth
- Hanusch Krankenhaus, Vienna, Austria
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - VITAZ, Sint-Niklaas
- Brazil (14):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - Upeclin - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu - UNESP, Botucatu
  - Hemocentro Unicamp, Campinas
  - Hospital Uopeccan - Centro de Pesquisa Clinica, Cascavel
  - Centro Integrado de Oncologia de Curitiba, Curitiba
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba
  - Instituto do Câncer - Hospital São Vicente de Paulo, Passo Fundo
  - Centro Gaucho Integrado - Mae de Deus Center, Porto Alegre
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Centro Integrado de Pesquisa Clinica, São José do Rio Preto
  - Hospital BP, São Paulo
  - Hospital da Clinicas da Faculdade de Medicina da USP, São Paulo
  - Hospital Santa Marcelina, São Paulo
- Canada (3):
  - Royal Victoria Hospital-Montreal, Montreal
  - Hopital de L'Enfant Jesus, Québec
  - Cancer Care Manitoba, Winnipeg
- Chile (4):
  - Inmunocel, Santiago
  - CeCim Biocinetic, Santiago
  - Sociedad de Investigaciones Médicas Limitada, Temuco
  - Centro de Investigaciones Clínicas Viña del Mar (CIC), Viña del Mar
- China (18):
  - The Second Xiangya Hospital of Central South University, Changsha
  - Hunan Cancer Hospital, Changsha
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Southern Medical University Nanfang Hospital, Guangzhou
  - Hainan General Hospital, Haikou
  - First Affiliated Hosp of College of Med, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The Second Hospital of Anhui Medical University, Hefei
  - Jiangxi Provincial Cancer Hospital, Nanchang
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - Blood Institute of the Chinese Academy of Medical science, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Wu Han Tongji Hospital, Wuhan
  - The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu
- Czechia (6):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni Nemocnice Plzen, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (10):
  - CHD Vendee, La Roche-sur-Yon
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier Universitaire (Limoges) (CHU DUPUYTREN 1), Limoges
  - CHU de Nantes - Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital de la Pitie Salpetriere, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de Pontchaillou, Rennes
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen, Rouen
  - CHRU De Tours, Tours
- Germany (4):
  - Gemeinschaftspraxis für Hämatologie und Onkologie (Gefos), Dortmund
  - Onkologische Gemeinschaftspraxis / BAG, Dresden
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Medizinische Klinik und Poliklinik 1, Dresden
  - Universitätsklinikum Ulm, Ulm
- Hungary (2):
  - Debreceni Egyetem Orvos-es Egészsegtudomanyi Centrum, Debrecen
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Unita Sanitaria Locale di Reggio Emilia, Reggio Emilia
- Japan (2):
  - Kumamoto University Hospital, Kumamoto
  - Yamagata University Hospital, Yamagata
- New Zealand (4):
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Momentum Clinical Research, Newtown
  - Middlemore Clinical Trials, Papatoetoe
- Poland (8):
  - KO-MED Centra Kliniczne, Biała Podlaska
  - Szpital Uniwersytecki nr 1 im. Antoniego Jurasza, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Klinika Hematoonkologii i Transplantacji Szpiku,Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - AIDPORT Sp. z o.o., Skórzewo
  - Uniwersytecki Szpital Kliniczny Klinika, Wroclaw
- South Korea (4):
  - Inje Univ Busan Paik Hospital, Busan
  - The Catholic University of Korea-Seoul St. Mary's Hospital, Seocho-Gu
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (13):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario Infanta Leonor-INTERNAL MED, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Costa Del Sol, Marbella
  - Clinica Universitaria De Navarra, Pamplona
  - Hospital De Navarra, Pamplona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
- Taiwan (4):
  - Chang Bing Show Chwan Memorial Hospital, Changhua
  - Chang Gung Memorial Hospital - Chiayi, Chiayi County
  - National Cheng-Kung Uni. Hosp., Tainan
  - Koo Foundation Sun Yan-Sen Cancer Center, Taipei
- Turkey (Türkiye) (7):
  - Gazi University Faculty of Medicine, Ankara
  - 9 Eylul University Hospital, Balçova
  - Ege Üniversitesi, Bornova
  - Istanbul University Istanbul Medicine Faculty, Faith
  - American Hospital, Istanbul
  - Acıbadem Maslak Hastanesi, Istanbul
  - Ankara University Medicine Hospital, Mamak
- United Kingdom (5):
  - Bristol Haematology and Oncology Centre, Bristol
  - Castle Hill Hospital, Cottingham
  - HOPE Centre, Leicester
  - St Bartholomew's Hospital, London
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Pirtobrutinib (LOXO-305) Versus Ibrutinib in Participants With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) (BRUIN-CLL-314) — https://trials.lilly.com/en-US/trial/334656